CLINICAL TRIAL: NCT05274581
Title: Evaluating Scanning Competence Following a Structured POCUS Training Program for General Practitioners - A Hybrid Effectiveness-implementation Study
Brief Title: General Practitioners' POCUS Competence Following Structured Training
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Camilla Aakjær Andersen, Assistant professor, MD, PhD, Aalborg University
Other Study IDs: ID 242-2
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Ultrasound; General Practice; Family Medicine; Education; Competence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Course participants: Course participants er general practitioners who have signed-up to participate in an ultrasound course
  Interventions: Other: A new type of ultrasound course

INTERVENTIONS:
Other: A new type of ultrasound course — All participants will receive the educational intervention. The educations intervention consists of three teaching seminars over three months, a curriculum of 10 point-of-care ultrasound applications, an online learning platform providing educational support before, during and after the teaching sessions.

SUMMARY:
The overarching aim of this study is to investigate whether a new educational point-of-care ultrasound course tailored for general practitioners working in office-based general practice can lead to scanning competence at the end of the training program (three months after baseline) and if scanning competence can be maintained six months after baseline.

DETAILED DESCRIPTION:
Type of study:

This is a hybrid effectiveness-implementation study . The investigators will test the effectiveness of a new type of point-of-care ultrasound course, tailored to meet the educational needs of office-based general practitioners, in a real-world setting while gathering information on its delivery and the implementation of the intervention.

Setting:

This study will be conducted in office-based general practice in Denmark with the educational sessions taking place at an ultrasound educational facility.

The intervention:

The ultrasound course consists of three teaching seminars over three months, a curriculum of 10 point-of-care ultrasound (POCUS) applications, an online learning platform providing educational support before, during and after the teaching sessions.

The online platform includes instruction videos demonstrating the performance of POCUS, suggestions for additional literature, flashcards training the recognition of pathology, participant assignments to support the development of skills, self-quizzes to focus attention of learning outcomes and specific actioncards for each of the 10 POCUS applications framing the examinations in the clinical context. In addition, the online platform gives participants access to webinars and communication with other participants and teachers. A detailed description of the educational elements in the ultrasound course can be found in the attached study protocol.

Data collection:

The primary outcomes are the Objective Structured Assessment of Ultrasound Skills (OSAUS) score scored three (outcome 1) and six months (outcome 2) after baseline.

The OSAUS assessment tool has been developed and validated as a generic tool for assessing scanning competence. The OSAUS scale consists of seven items: 'indication for the examination', 'applied knowledge of ultrasound equipment', 'image optimization', 'systematic examination', 'interpretation of images', 'documentation of the examination' and 'medical decision-making' and each item is rated using a provided five-point Likert-scale with descriptions of performance ranging from very poor (score = 1) to excellent (score = 5). All items are weighted equally, as high inter-item correlation have been found previously. Hence, for each scanning modality a total score from 7 to 35 points may be achieved.

On the third teaching seminar (three months after baseline) and again six months after baseline, participants will have their scanning competence assessed by external experts. These experts are blinded to the participants previous experience and learning process.

The experts will assess the participants by asking the following questions:

- In which clinical scenarios would you perform this POCUS examination (Item 1 in the OSAUS)

The experts will ask participants to demonstrate the POCUS examination (for maximum five minutes) to assess the following:

* Applied knowledge of the ultrasound equipment (Item 2 in the OSAUS)
* Image optimazation (Item 3 in the OSAUS)
* Systematic examination (Item 4 in the OSAUS)
* Interpretation of images (Item 5 in the OSAUS)

The experts will present the participants with two picture of common pathology and ask the participants the following questions:

* How would you interpret these ultrasound findings? (Item 5 in the OSAUS)
* If you were to describe this examination in the medical record, what would you write? (Item 6 in the OSAUS)
* What would you do if you found it? (Item 7 in the OSAUS) The OSAUS score will also be used for secondary outcomes S1, S2 and S3)

Immediately before each competence assessment by experts, participants will be asked to fill out a questionnaire where they declare whether or not they have POCUS scanning competence within this scanning modality to perform the scan un-supervised in general practice (outcomes 6 and 7). The expert assessor are blinded to this declaration.

In addition, the following process-related outcomes will be collected:

The GPs keep a log book of all scans they perform. The number of scans of the 10 POCUS modalities performed during months 1 to 3 and month 4 to 6 are summarized (outcome 8).

The GPs will register the number of adverse events and near-miss cases associated with their use of POCUS during months 1 to 6, in a questionnaire specifically designed for this purpose (outcome 9).

The GPs activity on the online platform will be registered during the educational period (months 1-3) (outcome 10).

Background characteristics of participating GPs At baseline the following participant characteristics will be collected: Age (years), gender (M, F, other), previous use of ultrasound (number of months with regular use), previous ultrasound courses of minimum 1 day duration (yes/no), scanner type (low range, mid range, high end), type of practice (collaboration, partnership, solo), location of practice (urban, rural, mixed), number of patients assigned to the practice, number of GPs working in the practice will be presented.

Data analysis:

All statistical analyses will be performed using STATA version 17 (StataCorp, Texas, USA) and analyzed according to a predefined statistical analysis plan, which will be uploaded prior to the data collection for the primary outcome (three months after baseline).

ELIGIBILITY:
Inclusion criteria:

1. GP, i.e., be a postgraduate medical doctor with a specialization in general practice.
2. Work in office-based general practice in Denmark
3. Have access to an ultrasound device in the practice during the study period

Exclusion criteria:

1. GPs with a possible conflict of interest (e.g., industry affiliation related to the use of ultrasound)
2. No signed informed consent to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Twenty GPs working in office-based general practice in Denmark, who have signed up for a PLO-e ultrasound course, will be invited to participate in the study. To participate a GPs must fulfill the inclusion criteria and not the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Participants' ultrasound competence score after three months | three months after baseline
  Participants' ultrasound competence score across ten scanning modalities (The Objective Structured Assessment of Ultrasound Skills (OSAUS)) after the educational period
Participants' ultrasound compentence score after six months | six months after baseline
  Participants' ultrasound competence score across ten scanning modalities (The Objective Structured Assessment of Ultrasound Skills (OSAUS)) six months after baseline

SECONDARY OUTCOMES:
Participants' ultrasound competence items scores | three months after baseline
  Participants' total ultrasound competence score (The Objective Structured Assessment of Ultrasound Skills (OSAUS) 7-35) and the item scores (1-5), for each of the ten scanning modalities included in the curriculum.
Participants' ultrasound compentence scores above avarage after three months | three months after baseline
  The proportion of participants, who have an ultrasound competence score (OSAUS score) of three or more, after the educational period, in all of the seven OSAUS items, for each of the ten scanning modalities included in the curriculum
Participants' ultrasound compentence scores above avarage after six months | six months after baseline
  The proportion of participants, who have an ultrasound competence score (OSAUS score) of three or more, in all of the seven OSAUS items, for each of the ten scanning modalities included in the curriculum
Participants' self-rated ultrasound compentence after three months | three months after baseline
  The proportion of participants, who rate themselves to be competent to perform un-supervised POCUS in general practice, after the educational period, for each of the ten scanning modalities included in the curriculum.
Participants' self-rated ultrasound compentence after six months | six months after baseline
  The proportion of participants, who rate themselves to be competent to perform un-supervised POCUS in general practice, six months after baseline, for each of the ten scanning modalities included in the curriculum.

OTHER OUTCOMES:
Number of performed POCUS examinations | months 1-6 after baseline
  The number of performed POCUS examinations by each participant in the first six months after introducing POCUS use in general practice
Number of adverse events and near-miss cases | months 1-6 after baseline
  The number of adverse events and near-miss cases associated with the use of POCUS reported by the participants in the first six months after introducing POCUS use in general practice
Participants' completion of educational elements | months 1-3 after baseline
  The proportion of participants, who have completed the different educational elements in the educational intervention three months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Camilla A Andersen, Principal Investigator — Aalborg University
Locations (1):
- Center for General Practice at Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
We aim to publish positive, negative or inconclusive results of the study in a peer-reviewed journal. The project group will also present results at conferences.

REFERENCES:
- [Derived] Andersen CA, Lundbye-Christensen S, Riis A, Mehnert U, Lokkegaard T, Mengel-Jorgensen T, Rasmussen LD, Soll N, Stork B, Andersen SK, Pil L, Stjernebjerg C, Graumann O, Jensen MB. General practitioners' scanning competence following tailored ultrasound training: a hybrid effectiveness-implementation study. BMC Med Educ. 2025 May 20;25(1):733. doi: 10.1186/s12909-025-07356-8. PMID 40394656

DOCUMENTS (2):
  • Study Protocol (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT05274581/Prot_002.pdf
  • Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT05274581/SAP_004.pdf